CLINICAL TRIAL: NCT07208331
Title: Evaluation of an Integrated, Digital, Nurse-led, Remote Monitoring Care Pathway for Cardiovascular Risk Management
Acronym: TELE-CVRM
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Cardiology Centres of the Netherlands (Unknown)
Responsible Party: Principal Investigator, M.M. Winter, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2025.0543
Record Dates: First submitted 2025-09-25; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Hypertension; Dyslipidemia
Keywords: Telemonitoring; Lipids; eHealth; Screening; Telemedicine; Risk factor management; Blood pressure
MeSH Terms: conditions — Atherosclerosis; Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the implementation of a structured, digital, nurse-led, remote monitoring care pathway for cardiovascular risk management (CVRM). Participants will receive this care as part of routine clinical practice. In addition to standard follow-up, participants will complete questionnaires on quality of life, medication adherence, system usability, and patient satisfaction.

DETAILED DESCRIPTION:
CVRM is essential for patients at increased risk of cardiovascular disease (CVD) as well as for those with established atherosclerotic cardiovascular disease (ASCVD). Monitoring blood pressure and lipid profiles is crucial to achieving guideline-recommended targets. However, many patients fail to reach these targets despite the availability of effective therapies, resulting in an increased risk of recurrent events. Meanwhile, the burden of CVD continues to rise, creating significant pressure on healthcare systems.

A digital care pathway may improve therapy adherence and outcomes by enabling personalized, data-driven care. This study evaluates the effectiveness of a nurse-led, telemonitoring pathway for CVRM in routine practice, where patients measure their blood pressure and LDL-c levels at home. The study aims to improve risk stratification, support earlier intervention, and optimize lipid and blood pressure control, ultimately leading to better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All patients enrolled in the program (high-risk and very high-risk patients)

Exclusion Criteria:

* Not able to provide informed consent
* No access to smartphone and/or tablet
* Inability to use digital tools required for the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in the digital CVRM program will be invited to participate in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients on-target for LDL-c | Baseline and 1 year
  Proportion of patients achieving guideline-recommended LDL-c targets

SECONDARY OUTCOMES:
Mean LDL-c | Baseline and 1 year follow-up
  The mean of LDL-c values in mmol/L, measured at-home
Number of patients achieving blood pressure control | Baseline and 1 year
  Proportion of patients achieving guideline-recommended blood pressure targets
Change in home-measured blood pressure values | Baseline and 1 year
  Change in blood pressure values measured at home with telemonitoring in mmHg
Number of medication changes | 1 year
  Changes in lipid-lowering and antihypertensive medications, defined as change in dose and change in medication type
5-item Medication Adherence Report Scale (MARS-5) | Baseline and 1 year
  5 questions about medication adherence, with higher scores indicating better adherence
Visual Analog Scale (VAS) for medication adherence | Baseline and 1 year
  The scale ranges from 0% to 100%, with higher scores indicating better medication adherence
Quality of life (QoL) | Baseline and 1 year
  Using the EuroQoL-5D questionnaire
Telehealth Usability Questionnaire (TUQ) | Baseline and 1 year
  18 questions on patient satisfaction and usability, with higher scores indicating better satisfaction
Hospitalization | 12 and 24 months
  Unplanned cardiovascular (re)hospitalization
MACE | 12 and 24 months
  Cardiovascular death, myocardial infarction, any documented stroke (ischemic or hemorrhagic), ischemia-driven revascularization
All-cause mortality | 12 and 24 months
  Total number of deaths from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Centers of the Netherlands (CCN), Amsterdam, North Holland, Netherlands